CLINICAL TRIAL: NCT04804540
Title: A Multicenter, Single-arm, Open-label, Phase 4 Study to Evaluate the Safety and Efficacy of Vedolizumab in Indian Patients With Ulcerative Colitis and Crohn's Disease
Brief Title: A Study of Vedolizumab in People With Ulcerative Colitis and Crohn's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vedolizumab-4020; EUPAS23702 (Other: ENCePP)
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Ulcerative Colitis; Crohn Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vedolizumab 300 mg (Experimental): Vedolizumab 300 mg IV infusion will be administered once in Weeks 0, 2 and 6 during induction phase and in Weeks 14, 22, 30, 38 and 46 during maintenance phase.
  Interventions: Drug: Vedolizumab IV

INTERVENTIONS:
Drug: Vedolizumab IV — Vedolizumab IV infusion
  Other Names: Kynteles

SUMMARY:
Vedolizumab is a medicine that helps to reduce inflammation and pain in the digestive system. In this study, people with ulcerative colitis or Crohn's disease will be treated with vedolizumab. The main aim of the study is to check for side effects from vedolizumab.

At the first visit, the study doctor will check who can take part. Participants will receive vedolizumab slowly through a vein (infusion). Participants will regularly visit the clinic for up to 46 weeks for more infusions of Vedolizumab. During these visits, the study doctor will check if there are any side effects from this treatment.

Participants will visit the clinic for a final check-up up to 16 weeks after their final infusion of Vedolizumab. Clinic staff will arrange a phone call 6 months after their final infusion of Vedolizumab for a further check-up.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab. Vedolizumab is being tested to treat people who have active UC or CD.

The study will enroll approximately 150 patients. Participants will be assigned to the vedolizumab treatment group.

•Vedolizumab 300 mg

Vedolizumab 300 mg IV infusion will be administered once in Weeks 0, 2, 6 and 10 (CD-participants who have not shown a response can receive a dose at Week 10) during induction phase and in Weeks 14, 22, 30, 38 and 46 during maintenance phase.

This multicentre trial will be conducted in India. The overall time to participate in this study is 74 weeks. Participants will make multiple visits to the clinic, and will be contacted by telephone plus a final visit after receiving their last dose of drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of moderately to severely active ulcerative colitis (UC) or Crohn's disease (CD) at least 3 months prior to screening, with a Full Mayo Score of 6-12 for UC and a Harvey Bradshaw Index (HBI) score of >=8 for CD at the time of enrolment.
2. Has demonstrated, an inadequate response to, loss of response to, or intolerance to at least 1 of the following agents:

   1. Conventional therapy
   2. TNF-α alpha antagonist

Exclusion Criteria:

1. Has undergone an ileostomy, colostomy, or has known fixed symptomatic stenosis of the intestine.
2. Has active or latent tuberculosis (TB).
3. Has had a prior exposure to vedolizumab or a history of hypersensitivity or allergies to vedolizumab, natalizumab, efalizumab, or rituximab.
4. Has a positive progressive multifocal leukoencephalopathy (PML) subjective symptom checklist during screening or prior to the administration of study drug on Day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (17):
- India (17):
  - Government General Hospital, Guntur, Andhra Pradesh
  - Institute of Gastroenterology and Liver Disease Dispur Hospitals, Guwahati, Assam
  - Indira Gandhi Institute of Medical Sciences, Patna, Bihar
  - Gastroplus Digestive Disease Centre Pvt.Ltd, Ahmedabad, Gujarat
  - Surat Institute of Digestive Sciences, Surat, Gujarat
  - Banglore Medical College & Research Institute, Bangalore, Karnatka
  - Midas Multispeciality Hospital, Nagpur, Maharashtra
  - Dr. Ram Manohar Lohia Hospita Hospital, New Delhi, National Capital Territory of Delhi
  - Maulana Azad Medical college & Associated G B Pant Hospital, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Dayanand Medical College and Hospital, Ludhiana, Punjab
  - VGM Hospital- Institute of Gastroenterology, Coimbatore, Tamil Nadu
  - Asian Institute of Gastroenterology, Hyderabad, Telangana
  - Yashoda Hospitals, Secunderabad, Telangana
  - King George's Medical University, Lucknow, Uttar Pradesh
  - Osmania General Hospital, Hyderabad
  - Deccan College of Medical Sciences, Hyderabad

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Related Info — https://clinicaltrials.takeda.com/study-detail/5f6b60394db2bf003ab4a247

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at the 17 investigative sites in India from 08 December 2021 to 02 February 2024.
Pre-assignment Details: A total of 150 participants diagnosed with moderate to severe Ulcerative Colitis (UC) (102 participants) and Crohn's Disease (CD) (48 participants) were enrolled to receive vedolizumab treatment in this study.
Groups:
- UC Participants: Vedolizumab 300 mg: Participants received vedolizumab 300 milligrams (mg), intravenous (IV) infusion, once at Weeks 0, 2, 6, 14, 22, 30, 38 and 46.
- CD Participants: Vedolizumab 300 mg: Participants received vedolizumab 300 mg, IV infusion, once at Weeks 0, 2, 6, 10 14, 22, 30, 38 and 46.
Period: Overall Study
Arm/Group | UC Participants: Vedolizumab 300 mg | CD Participants: Vedolizumab 300 mg
Started | 102 | 48
Completed | 76 | 35
Not Completed | 26 | 13
Not completed — Adverse Event | 26 | 13

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAS) included all enrolled participants who received at least 1 dose of study drug.
Groups:
- UC Participants: Vedolizumab 300 mg: Participants received vedolizumab 300 mg, IV infusion, once at Weeks 0, 2, 6, 14, 22, 30, 38 and 46.
- Total: Total of all reporting groups
Arm/Group | UC Participants: Vedolizumab 300 mg | CD Participants: Vedolizumab 300 mg | Total
Number analyzed (Participants) | 102 | 48 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.55 (11.190) | 32.60 (10.849) | 36.65 (11.391)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 32 | 67
  Male | 67 | 16 | 83
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Indian | 102 | 48 | 150

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs)
Description: AE was defined as any untoward medical occurrence in clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with the treatment. AE can therefore be any unfavourable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with use of a drug, whether or not it is considered related to the drug. A SAE was any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of an existing hospitalization, resulted in significant disability or incapacity, was a congenital anomaly/birth defect or was a medically important event. An AESI (serious or nonserious) was one of scientific and medical concern specific to the compound or program.
Time Frame: From first dose of study drug up to 24 weeks after the last dose (up to 70 weeks)
Population: SAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | UC Participants: Vedolizumab 300 mg | CD Participants: Vedolizumab 300 mg
Number analyzed (Participants) | 102 | 48
Participants
  Participants with AEs | 54 | 29
  Participants with SAEs | 6 | 2
  Participants with AESIs | 4 | 0

2. Primary Outcome: Number of Participants With Adverse Drug Reactions (ADRs) and Unexpected ADRs
Description: An ADR was an AE for which there was at least a reasonable suspicion of a causal relationship between an AE and a suspected medicinal product. An unexpected ADR was an ADR with the nature, severity, or outcome which was not consistent with the product insert.
Time Frame: From first dose of study drug up to 24 weeks after the last dose (up to 70 weeks)
Population: SAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | UC Participants: Vedolizumab 300 mg | CD Participants: Vedolizumab 300 mg
Number analyzed (Participants) | 102 | 48
Participants
  Participants with ADRs | 5 | 0
  Participants with Unexpected ADRs | 2 | 0

3. Secondary Outcome: Percentage of UC Participants With Clinical Response at Weeks 14, 30 and 46
Description: Clinical response for UC participants was defined as decrease in Simple Clinical Colitis Activity Index (SCCAI) of greater than and equal to (>=) 3 from baseline or by physician assessment of clinical response. The SCCAI consists of five colitis activity symptom items (bowel frequency per day, bowel frequency per night, urgency of defecation, blood in stool, and general well-being) along with an assessment of extracolonic manifestations. Bowel frequency per night is scored on a 0-2 scale and General well-being is scored on a 0-4 scale. The other 3 symptom scores are scored on a 0-3 scale. 1 point each is added for the presence of any extracolonic manifestation (i.e., arthritis, erythema nodosum, pyoderma gangrenosum, and uveitis). The total overall possible scoring range was 0-19 with increasing scores being indicative of more colitis activity.
Time Frame: At Weeks 14, 30 and 46
Population: SAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UC Participants: Vedolizumab 300 mg
Number analyzed (Participants) | 102
percentage of participants
  At Week 14 | 54.9 [44.7 to 64.8]
  At Week 30 | 62.7 [52.6 to 72.1]
  At Week 46 | 73.5 [63.9 to 81.8]

4. Secondary Outcome: Percentage of CD Participants With Clinical Response at Weeks 14, 30 and 46
Description: Clinical response for CD participants was defined as decrease in Harvey Bradshaw Index (HBI) of >= 3 points from baseline. HBI was composed of five clinical parameters: general well-being (0-4, where higher score means lower wellbeing), abdominal pain (0-3, higher score means more severe pain), number of liquid stools/day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score was the sum of individual parameters. The score ranged from a minimum score of 0 to no pre-specified maximum score as it depended on the number of liquid stools, where higher scores indicated more severe disease. The score < 5 is considered as clinical remission, 5-7 mild, 8-16 moderate, and >16 severe disease. A higher score indicated a worse outcome.
Time Frame: At Weeks 14, 30 and 46
Population: SAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CD Participants: Vedolizumab 300 mg
Number analyzed (Participants) | 48
percentage of participants
  At Week 14 | 72.9 [58.2 to 84.7]
  At Week 30 | 70.8 [55.9 to 83.0]
  At Week 46 | 68.8 [53.7 to 81.3]

5. Secondary Outcome: Percentage of UC Participants With Clinical Remission at Weeks 14, 30 and 46
Description: Clinical remission for UC participants was defined as decrease in SCCAI of less than and equal to (<=) 2 with no individual score > 1. The SCCAI consists of five colitis activity symptom items (bowel frequency per day, bowel frequency per night, urgency of defecation, blood in stool, and general well-being) along with an assessment of extracolonic manifestations. Bowel frequency per night is scored on a 0-2 scale and General well-being is scored on a 0-4 scale. The other 3 symptom scores are scored on a 0-3 scale. 1 point each is added for the presence of any extracolonic manifestation (i.e., arthritis, erythema nodosum, pyoderma gangrenosum, and uveitis). The total overall possible scoring range was 0-19 with increasing scores being indicative of more colitis activity.
Time Frame: At Weeks 14, 30 and 46
Population: SAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UC Participants: Vedolizumab 300 mg
Number analyzed (Participants) | 102
percentage of participants
  At Week 14 | 39.2 [29.7 to 49.4]
  At Week 30 | 43.1 [33.4 to 53.3]
  At Week 46 | 52.0 [41.8 to 62.0]

6. Secondary Outcome: Percentage of CD Participants With Clinical Remission at Weeks 14, 30 and 46
Description: Clinical remission for CD participants was defined as HBI of <= 4. HBI was composed of five clinical parameters: general well-being (0-4, where higher score means lower wellbeing), abdominal pain (0-3, higher score means more severe pain), number of liquid stools/day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score was the sum of individual parameters. The score ranged from a minimum score of 0 to no pre-specified maximum score as it depended on the number of liquid stools, where higher scores indicated more severe disease. The score < 5 is considered as clinical remission, 5-7 mild, 8-16 moderate, and >16 severe disease. A higher score indicated a worse outcome.
Time Frame: At Weeks 14, 30 and 46
Population: SAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CD Participants: Vedolizumab 300 mg
Number analyzed (Participants) | 48
percentage of participants
  At Week 14 | 47.9 [33.3 to 62.8]
  At Week 30 | 45.8 [31.4 to 60.8]
  At Week 46 | 56.3 [41.2 to 70.5]

7. Secondary Outcome: Percentage of UC and CD Participants Who Discontinued Vedolizumab
Description: Vedolizumab discontinuation was defined as ceasing vedolizumab, or a treatment gap >= 90 days between consecutive doses.
Time Frame: From first dose of study drug up to Week 46
Population: SAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UC Participants: Vedolizumab 300 mg | CD Participants: Vedolizumab 300 mg
Number analyzed (Participants) | 102 | 48
percentage of participants | 25.5 [17.4 to 35.1] | 27.1 [15.3 to 41.8]

8. Secondary Outcome: Percentage of UC Participants With Mucosal Healing at Week 46
Description: Mucosal healing was based on endoscopic evidence of no inflammation and healing of the mucosa as defined by a Mayo endoscopic sub-score of <=1 point. Full Mayo Score evaluated ulcerative colitis stage, based on four parameters: stool frequency, rectal bleeding, endoscopic evaluation, and Physician's global assessment. Each parameter of the score (including Mayo endoscopic sub-score) ranged from 0 (normal or inactive disease) to 3 (severe activity) yielding a total score of 0-12. The scores 0-2 were considered as clinical remission, 3-5 mild, 6-10 moderate, and 11-12 severe, with higher scores indicated more severe disease.
Time Frame: At Week 46
Population: SAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UC Participants: Vedolizumab 300 mg
Number analyzed (Participants) | 102
percentage of participants | 22.5 [14.9 to 31.9]

9. Secondary Outcome: Percentage of CD Participants With Mucosal Healing at Week 46
Description: Mucosal healing was based on endoscopic evidence of no inflammation and healing of the mucosa as defined by a Simple Endoscopic Score for Crohn Disease (SES-CD) 0-2 or SES-CD <=4 and at least a 2-point reduction from baseline with no sub-score >1. SES-CD assessed the size of mucosal ulcers, ulcerated surface, endoscopic extension, and the presence and type of narrowings. Each of the four SES-CD variables was scored from 0 to 3, with the sum of scores for each variable ranging from 0 to 15 yielding a total SES-CD score of 0-60, where higher scores indicated more severe disease.
Time Frame: At Week 46
Population: SAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CD Participants: Vedolizumab 300 mg
Number analyzed (Participants) | 48
percentage of participants | 8.3 [2.3 to 20.0]

10. Secondary Outcome: Percentage of UC Participants With Endoscopic Response at Week 46
Description: Endoscopic response was defined as decrease in Mayo endoscopic sub-score of >=1 point in UC participants. Full Mayo Score evaluated ulcerative colitis stage, based on four parameters: stool frequency, rectal bleeding, endoscopic evaluation, and Physician's global assessment. Each parameter of the score (including Mayo endoscopic sub-score) ranges from 0 (normal or inactive disease) to 3 (severe activity) yielding a total score of 0-12. The scores 0-2 are considered as clinical remission, 3-5 mild, 6-10 moderate, and 11-12 severe, where higher scores indicated more severe disease.
Time Frame: At Week 46
Population: SAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UC Participants: Vedolizumab 300 mg
Number analyzed (Participants) | 102
percentage of participants | 21.6 [14.0 to 30.8]

11. Secondary Outcome: Percentage of CD Participants With Endoscopic Response at Week 46
Description: Endoscopic response was defined as > 50% decrease in SES-CD in CD participants. SES-CD assessed the size of mucosal ulcers, ulcerated surface, endoscopic extension, and the presence and type of narrowings. Each of the four SES-CD variables was scored from 0 to 3, with the sum of scores for each variable ranged from 0 to 15 yielding a total SES-CD score of 0-60, where higher scores indicated more severe disease.
Time Frame: At Week 46
Population: SAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CD Participants: Vedolizumab 300 mg
Number analyzed (Participants) | 48
percentage of participants | 12.5 [4.7 to 25.2]

12. Secondary Outcome: Change From Baseline in Patient-reported Quality of Life (Short Inflammatory Bowel Disease Questionnaire [SIBDQ]) Scores at Weeks 14, 30, and 46
Description: The SIBDQ was a valid and reliable instrument used to assess quality of life in adult participants with Inflammatory Bowel Disease (IBD). It was a 10-item questionnaire that included questions on 4 domains of health-related quality of life (HRQoL): bowel systems, emotional function, social function, and systemic function and was scored on a 7-point Likert scale from 1 (severe problem) to 7 (no problems at all). A total SIBDQ score was calculated by summing the scores from each domain; the total SIBDQ score ranged from 10 (poor HRQoL) to 70 (optimum HRQoL). Higher values of SIBDQ represented a better quality of life.
Time Frame: Baseline, Weeks 14, 30 and 46
Population: SAS included all enrolled participants who received at least 1 dose of study drug. Here, "overall number of participants analyzed" signified participants who were evaluable for this outcome measure and "number analyzed" signified participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UC Participants: Vedolizumab 300 mg | CD Participants: Vedolizumab 300 mg
Number analyzed (Participants) | 91 | 45
score on a scale
  Change at Week 14 | 8.4 (12.91) | 8.3 (12.24)
  Change at Week 30: number analyzed (Participants) | 81 | 42
  Change at Week 30 | 12.9 (13.16) | 8.4 (14.31)
  Change at Week 46: number analyzed (Participants) | 81 | 37
  Change at Week 46 | 13.0 (12.84) | 10.6 (15.91)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 24 weeks after the last dose (up to 70 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | UC Participants: Vedolizumab 300 mg | CD Participants: Vedolizumab 300 mg
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/48
Serious Adverse Events (participants affected / at risk) | 6/102 | 2/48
Other Adverse Events (participants affected / at risk) | 25/102 | 19/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UC Participants: Vedolizumab 300 mg (N=102) | CD Participants: Vedolizumab 300 mg (N=48)
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Tuberculous pleurisy (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UC Participants: Vedolizumab 300 mg (N=102) | CD Participants: Vedolizumab 300 mg (N=48)
Anaemia (Blood and lymphatic system disorders) | 8 | 6
Aphthous ulcer (Gastrointestinal disorders) | 0 | 3
Colitis ulcerative (Gastrointestinal disorders) | 7 | 0
Dizziness (Nervous system disorders) | 3 | 3
Headache (Nervous system disorders) | 5 | 4
Pyrexia (General disorders) | 7 | 6
Vomiting (Gastrointestinal disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT04804540/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT04804540/SAP_001.pdf